CLINICAL TRIAL: NCT02952768
Title: The Novel US-C-A-B Protocol: Curriculum Implementation and Evaluation of Proficiency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 201505089RINA
Record Dates: First submitted 2016-10-26; First posted 2016-11-02 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2016-10

CONDITIONS: Ultrasound Therapy; Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ultrasound training (Other): The aims were to develop a novel, resuscitative ultrasound-circulation-airway-breathing (US-C-A-B) protocol, to implement a short curriculum for ultrasound training and to assess the feasibility.
  Interventions: Behavioral: ultrasound training

INTERVENTIONS:
Behavioral: ultrasound training — Through the ultrasound-circulation-airway-breathing training curriculum to integrate the ultrasound into clinical practice.

SUMMARY:
Ultrasound is a frequently used diagnostic tool in the emergency department and suggested to have a role during resuscitation. The aims of this study were to develop a novel, resuscitative ultrasound-circulation-airway-breathing (US-C-A-B) protocol, to implement a short curriculum and to assess the feasibility.

The US-C-A-B protocol was built in an advanced life support-compliant manner. It involved a 3-part assessment: (1) C: subxiphoid 4-chamber view of the heart; (2) A: tracheal ultrasound; and (3) B: bilateral lung sliding. It could be used for direct confirmation for the C-A-B and searching the possible cause of cardiac arrest.

A half-day curriculum was designed, and comprised of one-hour didactics and 3-hour small-group hand-on training. Assessments were performed, including a written test, the US image acquisition and a satisfaction survey. From August 1, 2014 to March 31, 2016, the multi-center emergency physicians who attended the US-C-A-B curricula were enrolled prospectively.

DETAILED DESCRIPTION:
Ultrasound is a frequently used diagnostic tool in the emergency department and suggested to have a role during resuscitation. The aims of this study were to develop a novel, resuscitative ultrasound-circulation-airway-breathing (US-C-A-B) protocol, to implement a short curriculum and to assess the feasibility.

The US-C-A-B protocol was built in an advanced life support-compliant manner. It involved a 3-part assessment: (1) C: subxiphoid 4-chamber view of the heart; (2) A: tracheal ultrasound; and (3) B: bilateral lung sliding. It could be used for direct confirmation for the C-A-B and searching the possible cause of

ELIGIBILITY:
Inclusion Criteria:

* The enrolled participants were emergency physicians of the National Taiwan University Hospital (NTUH), the Far-Eastern Memorial Hospital (FEMH) and the Chang-Kung Memorial Hospital (CKMH), three teaching hospitals in Taiwan.

Exclusion Criteria:

* Not emergency physicians.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-08; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The time of the US image acquisition | 6 months
  The 6-month evaluation was performed in cardiac arrest patients. The ultrasound operation time was from the time to initiate the ultrasound exam to when the sonographers to inteprete the results, using the ultrasound recorder.

SECONDARY OUTCOMES:
Learning efficacy was assessed with a written test with 10 multi-choice questions. | through study completion, an average of 1 year
  The written test with 10 multi-choice questions, including ALS knowledge, and still US image interpretation of C-A-B was performed before and after completion of the course.
A satisfaction survey with a 5-point Likert scale. | through study completion, an average of 1 year
  The post-course satisfaction survey queried the participants in regards to educational value, knowledge acquisition and self-confidence at the end of the course. The survey consisted of 5 items, using a 5-point Likert scale.
The time of the US image acquisition | through study completion, an average of 1 year
  The participants were asked for to produce adequate views of each C-A-B category and consecutive C-A-B exams in the same live model after completion, recorded by the DVD recorder. The time to achieve the views was measured from positioning of the probe on the skin to maintaining an adequate image for at least 3 seconds. The videos were edited that the faces of the participants were covered, and reviewed blindly and independently by the authors. The 6-month evaluation was performed in cardiac arrest patients. The ultrasound operation time was from the time to initiate the ultrasound exam to when the sonographers to inteprete the results, using the ultrasound recorder.

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Ching Lien, Ph.D., Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No